CLINICAL TRIAL: NCT06938503
Title: A Prospective, Single-Arm Study of Nab-paclitaxel/Gemcitabine Combined With Nimotuzumab Sequential Irreversible Electroporation Ablation for Locally Advanced Pancreatic Cancer
Brief Title: AG Plus Nimotuzumab Sequential Irreversible Electroporation Ablation for Locally Advanced Pancreatic Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IST-PC-202501
Record Dates: First submitted 2025-04-14; First posted 2025-04-22 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: Pancreatic Cancer, Adult
MeSH Terms: conditions — Pancreatic cancer, adult | interventions — nimotuzumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AG+Nimotuzumab (Experimental)
  Interventions: Drug: AG regimen; Drug: Nimotuzumab

INTERVENTIONS:
Drug: AG regimen — Patients will receive 4 cycles of AG (gemcitabine 1000 mg/m^2 and nab-paclitaxel 125 mg/m^2 on days 1 and 8 of a 21-day cycle), followed by Irreversible Electroporation Ablation and 3 cycles of adjuvant AG (gemcitabine 1000 mg/m^2 and nab-paclitaxel 125 mg/m^2 on days 1 and 8 of a 21-day cycle).
Drug: Nimotuzumab — Patients will receive 4 cycles of Nimotuzumab (400 mg on days 1, 8, and 15 of a 21-day cycle), followed by Irreversible Electroporation Ablation and 3 cycles of adjuvant Nimotuzumab (400 mg on days 1, 8, and 15 of a 21-day cycle).

SUMMARY:
This is a prospective, open-label, single arm clinical study. The main purpose of the study is to evaluate the clinical efficacy and safety of nab-paclitaxel/gemcitabine combined with nimotuzumab sequential irreversible electroporation ablation for locally advanced pancreatic cancer. The main endpoint is overall survival (OS).

DETAILED DESCRIPTION:
This clinical study is designed as a prospective, open-label, single arm study to evaluate the clinical efficacy and safety of nab-paclitaxel/gemcitabine combined with nimotuzumab sequential irreversible electroporation ablation for locally advanced pancreatic cancer. This study is divided into two stages: in stage I, all patients will receive 4 cycles of nab-paclitaxel/gemcitabine (AG regimen, 3 weeks as a cycle) and nimotuzumab. Imaging reexamination will be conducted 12 weeks later. In stage II, patients who are without disease progression (PD) will receive irreversible electroporation ablation and at least 3 cycles of adjuvant treatment (AG and nimotuzumab). If the imaging evaluation shows disease progression (PD), then the subsequent treatment will be changed to the standard treatment in hospital. The main endpoint is overall survival (OS). Additional end points included progression-free survival (PFS), objective response rate (ORR), disease control rate (DCR), safety, etc.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age 18-75 years old, gender unlimited;
* 2. Histologically or cytologically confirmed pancreatic cancer;
* 3. Confirmed as locally advanced pancreatic cancer by CT/MRI imaging, with no evidence of distant metastasis;
* 4. No prior chemotherapy or other tumor systemic therapy;
* 5. Measurable disease according to RECIST criteria v1.1;
* 6. Adequate organ and bone marrow function, defined as follows: hemoglobin≥9.0 g/dL; absolute neutrophil count (ANC)≥1.5×10^9/L; platelets≥100×10^9/L; serum total bilirubin (TBIL)≤1.5×ULN; aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 times the upper limit of normal (ULN); serum creatinine≤1.5×ULN or estimated creatinine clearance > 60 mL/min;
* 7. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 2;
* 8. Life expectancy is expected to be ≥3 months;
* 9. Fertile subjects are willing to take contraceptive measures during the study period.
* 10. Good compliance and signed informed consent voluntarily.

Exclusion Criteria:

* 1. Refuse chemotherapy or surgery;
* 2. Other part (e.g. peritoneum, lung, bone, brain) metastasis;
* 3. History of other malignancies (except cured basal cell carcinoma of the skin and carcinoma in situ of the cervix);
* 4. Accompanied by other serious diseases, including but not limited to: compensatory heart failure (NYHA grade III and IV), unstable angina, poorly controlled arrhythmias, uncontrolled hypertension (SBP>160mmHg or DBP>100mmHg); active infections; unmanageable diabetes mellitus; presence of uncontrolled pleural effusion, pericardial effusion, or ascites requiring drainage; severe portal hypertension; gastric outlet obstruction; Respiratory insufficiency;
* 5. Undergone major surgery within 30 days;
* 6. Participated in other drug related clinical trials within 4 weeks;
* 7. Known allergy to prescription or any component of the prescription used in this study;
* 8. With HIV, or active hepatitis (hepatitis B, hepatitis C);
* 9. Failure to recover from treatment-related toxicity to ≤ grade 1 (adverse events such as alopecia judged by the researcher not to affect the treatment with the research drug are excluded);
* 10.Other reasons that are not suitable to participate in this study according to the researcher's judgment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-04-21 (Estimated); Primary Completion 2028-04-25 (Estimated); Study Completion 2028-04-28 (Estimated)

PRIMARY OUTCOMES:
overall survival (OS) | Up to 24 months
  OS, defined as the time from the beginning of treatment to death due to any cause.

SECONDARY OUTCOMES:
progression-free survival (PFS) | Up to 24 months
  PFS, defined as the time from the beginning of treatment to disease progression or all-cause death. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Objective response rate (ORR) | Up to 24 months
  Objective response rate (ORR), including complete response (CR) and partial response (PR). Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by CT/MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), at least a 30% decrease in the sum of the longest diameter of target lesions.
Disease control rate (DCR) | Up to 24 months
  Disease control rate (DCR), including complete response (CR) and partial response (PR) and stable disease(SD). Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by CT/MRI: CR, disappearance of all target lesions; PR, at least a 30% decrease in the sum of the longest diameter of target lesions. SD, neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD (PD, defined as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions).